CLINICAL TRIAL: NCT01324921
Title: Effect of Nutritional Products on Metabolic Parameters in Subjects With Type 2 Diabetics
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Bobbie Swearengin, Director Clinical Research Operations, Abbott Nutrition
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BK40
Record Dates: First submitted 2011-03-27; First posted 2011-03-29 (Estimated); Last update posted 2011-03-30 (Estimated); Status verified 2011-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Breakfast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- No breakfast/beverage only (Placebo Comparator): 12 fluid ounces made up of one of some combination of the following: decaffeinated coffee, decaffeinated tea or water, with non-nutritive sweetener
  Interventions: Other: No breakfast/beverage only
- Breakfast (Active Comparator): 1 serving of unflavored instant oatmeal and 12 fluid ounces made up of one of some combination of the following: decaffeinated coffee, decaffeinated tea or water, with non-nutritive sweetener
  Interventions: Other: Breakfast
- 10004RF (Experimental): 1 serving (8 fluid ounces) of the experimental beverage and 4 fluid ounces made up of one of some combination of the following: decaffeinated coffee, decaffeinated tea or water, with non-nutritive sweetener
  Interventions: Other: 10004RF

INTERVENTIONS:
Other: No breakfast/beverage only — 12 fluid ounces made up of one of some combination of the following: decaffeinated coffee, decaffeinated tea or water, with non-nutritive sweetener
  Arms: No breakfast/beverage only
Other: Breakfast — 1 serving of unflavored instant oatmeal and 12 fluid ounces made up of one of some combination of the following:decaffeinated coffee, decaffeinated tea or water, with non-nutritive sweetener
  Arms: Breakfast
Other: 10004RF — 1 serving (8 fluid ounces) of the experimental beverage and 4 fluid ounces made up of one of some combination of the following:decaffeinated coffee, decaffeinated tea or water, with non-nutritive sweetener
  Arms: 10004RF

SUMMARY:
To compare the postprandial glycemic and insulinemic response of subjects with type 2 diabetes consuming a typical breakfast meal or no breakfast to 10004RF via a meal tolerance test (MTT).

ELIGIBILITY:
Inclusion Criteria:

1. type 2 diabetes
2. between 21 and 75 years of age
3. male or a non-pregnant, non-lactating female, at least 6 weeks postpartum or postmenopausal or surgically sterile
4. BMI is > 18.5 kg/m2 and <35 kg/m2
5. If subject is on a chronic medication such as an anti-hypertensive, lipid-lowering, thyroid medication or hormone therapy, they have been on constant dosage for at least two months prior to screening visit.

Exclusion Criteria:

1. Hemoglobin A1c value at screening of greater than or equal to 9%.
2. Uses exogenous insulin or exenatide for glucose control.
3. type 1 diabetes.
4. history of diabetic ketoacidosis.
5. current infection; has had inpatient surgery, or corticosteroid treatment in the last 3 months or antibiotics in the last 3 weeks prior to screening visit.
6. active malignancy
7. significant cardiovascular event ≤ six months prior to screening visit; or stated history of congestive heart failure.
8. end-stage organ failure or is status post organ transplant.
9. history of renal disease.
10. current hepatic disease.
11. history of severe gastroparesis.
12. chronic, contagious, infectious disease
13. taking any herbals, dietary supplements, or medications, other than anti-hyperglycemic medications, that could profoundly affect blood glucose.
14. clotting or bleeding disorders
15. allergic or intolerant to any ingredient found in the study products.
16. habitual user of tobacco products (

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Positive AUC for plasma glucose concentration | 0 to 180 minutes

SECONDARY OUTCOMES:
Plasma glucose concentrations | 0 to 180 minutes
Positive AUC for serum insulin concentration | 0-180 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Amy Devitt-Maicher, PhD, Study Chair — Abbott Nutrition
Locations (2):
- United States (2):
  - Provident Clinical Research and Consulting LLC, Glen Ellyn, Illinois
  - Radiant Research, Cincinnati, Ohio

REFERENCES:
- [Derived] Lohner S, Kuellenberg de Gaudry D, Toews I, Ferenci T, Meerpohl JJ. Non-nutritive sweeteners for diabetes mellitus. Cochrane Database Syst Rev. 2020 May 25;5(5):CD012885. doi: 10.1002/14651858.CD012885.pub2. PMID 32449201